CLINICAL TRIAL: NCT04566640
Title: Evolution of Fecal Incontinence in Patients With Rectal Static Disorder
Brief Title: Fecal Incontinence and Rectal Static Disorder
Acronym: NATUROSTATIQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_3074_NATUROSTATIQ
Record Dates: First submitted 2020-09-15; First posted 2020-09-28 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Fecal Continence Disorders; Posterior Pelvic Static Disorders
Keywords: Fecal incontinence; pelvic static disorders
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluate the rate of occurrence of fecal incontinence in patients who had surgery for posterior pelvic static disorder versus those with medical management.

The aim is also to assess the natural history of constipation symptoms and quality of life in patients with posterior pelvic static disorder.

DETAILED DESCRIPTION:
Data of all patients with posterior pelvic static disorder are collected prospectively and consecutively in the Fondamentum database since 2005, secured and hosted by the Rennes University Hospital.

The data from initial functional assessment, carried out as part of routine care between 2005 and 2019, include a clinical examination of pelvic static disorders, anorectal manometry, defecography, collection of symptoms by questioning and by a systematic questionnaire completed by the patient during the routine care consultation.

Patients identified from this database and meeting the selection criteria will receive an information letter along with a questionnaire and a stamped envelope for returning the questionnaire. The self-questionnaires will focus on collecting symptoms related to static disorders (incontinence, constipation, quality of life). Regarding the management of pelvic static disorder, we will detail whether it was operated or not, and what were the proposed medical care.

Upon receipt of the questionnaire, the new data will be entered into the research-specific database and will complete the clinical data resulting from the extraction of the care base The self-administered questionnaire sent to patients includes validated constipation (score of kess) and fecal incontinence (Cleveland) questionnaires, and quality of life questions from the validated SF36 questionnaire. It also includes a visual scale ranging from -5 to +5.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Having a disorder of posterior pelvic statics
* Diagnosed during the period 2005 - 2019
* Having a functional assessment in proctology between 2005 and 2019 in the proctology department of the Rennes University Hospital Center (CHU)
* This complete functional assessment was carried out in consultation with proctology, as part of routine care, and included :

  * Data from the interrogation
  * Reported symptoms: incontinence, constipation and quality of life (collected through questioning and through a questionnaire systematically completed by the patient during the routine care consultation),
  * A clinical examination
  * Anorectal manometry
  * A defecography
* no one who does not object to participation in the research

Exclusion Criteria:

* persons of full age subject to legal protection (safeguard of justice, guardianship, trusteeship), persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a posterior pelvic static disorder diagnosed and having benefited from a functional review in proctology between 2005 and 2019 in the proctology department of the University Hospital of Rennes
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Fecal incontinence defined by a Cleveland score > 5 | 6 weeks
  The objective of the study is to compare the rate of occurrence of fecal incontinence in patients who have had surgery for a disorder of posterior pelvic statics versus those with medical management.

SECONDARY OUTCOMES:
natural history of constipation symptoms in patients with posterior pelvic static disorders | 6 weeks
  Evaluation of Constipation Symptoms (Kess Score),
quality of life in patients with posterior pelvic static disorders | 6 weeks
  Quality of Life Score (Score SF36)

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided